CLINICAL TRIAL: NCT07062094
Title: Safety and Effectiveness of Orbera365™ Intragastric Balloon System: A Multi-Center, Prospective, Standard of Care Registry
Brief Title: Safety and Effectiveness of Orbera365™ Intragastric Balloon System
Acronym: Orbera365
Status: Not yet recruiting | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: E7235
Record Dates: First submitted 2025-06-24; First posted 2025-07-14 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Obesity
Keywords: Orbera365; Intragastric Balloon; Obesity; Orbera365™ IGB System
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 13 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Intragastric Balloon — The Orbera365™ IGB System is to be used in conjunction with a long-term supervised diet and behavior modification program designed to increase the possibility of long-term weight loss maintenance. The IGB is placed in the stomach and filled with sterile saline, causing it to expand into a spherical shape. The filled IGB is designed to occupy space and move freely within the stomach, potentially altering appetite and satiety to achieve weight loss.

SUMMARY:
This is a prospective, multi-center, standard of care registry offered to subjects in the EU only that have already agreed to receive the Orbera365™ Intragastric Balloon (IGB) System for weight loss. Subjects that agree to participate in the registry will have data reported associated with standard of care weight management visits during the time the device is implanted (in-dwell period), with an additional visit 30 days after the removal procedure.

DETAILED DESCRIPTION:
The study's objective is to confirm the safety of the Orbera365™ Intragastric Balloon (IGB) for extended in situ dwell time (from 6 months up to 12 months). This information can be collected from standard-of-care data. Up to ten (10) sites located in Europe are planned to participate in this registry. A minimum of 100 subjects are required for the registry. A maximum of 200 subjects may be enrolled into the registry.

The study population will include Obese patients ((Body Mass Index (BMI) 30-50 kg/m2)) who have already consented to receive the Orbera365™ IGB System, who previously failed to achieve and maintain weight loss with a supervised weight-control program.

Study subjects will also include obese and super obese patients (BMI 40 kg/m2 and above or a BMI of 35 kg/m2 with comorbidities) prior to obesity or other surgery, in order to reduce surgical risk.

The duration of study participation is expected to be up to thirteen months from study placement procedure. The total treatment with the study device will be no more than 12 months from placement. A 30-day post-removal assessment will be performed following the study removal procedure. The subject will have completed the study upon the completion of the 30-day post-removal assessment, regardless of when the study removal procedure occurred.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥ 18 years of age
2. Subject meets the indicated population for the device according to the Instructions for Use (IFU) including obese patients with the BMI of 30-50 kg/m2 for weight loss and patients with BMI 40 kg/m2 and above or a BMI of 35 kg/m2 with comorbidities before obesity or another surgery, unless contraindicated.
3. Subject is able to read, understand, and sign a written Informed Consent Form to participate in the registry

Exclusion Criteria:

1. Subject is planning on becoming pregnant during the one year following study device placement
2. Subject will complete follow-up visits at a location that the treating physician does not practice
3. Subjects who are unable or unwilling to take prescribed proton pump inhibitor medication for the duration of the device implant.
4. Current use or use within the three months before the baseline visit of over-the-counter or prescribed weight loss supplements/medications.
5. Subjects who have conditions that are contraindicated for Orbera365™ IGB System as per the IFU, including, but not limited to:

   * The presence of more than one IGB at the same time.
   * Any inflammatory disease of the gastrointestinal tract including esophagitis, gastric ulceration, duodenal ulceration, cancer or specific inflammation such as Crohn's disease
   * Potential upper gastrointestinal bleeding conditions
   * A large hiatal hernia of > 5cm or a hernia ≤ 5 cm associated with severe or intractable gastro- esophageal reflux symptoms
   * A structural abnormality in the esophagus or pharynx such as a stricture or diverticulum that could impede passage of the delivery catheter and/or an endoscope
   * Achalasia, symptoms suggestive of delayed gastric emptying, or presence of any other severe motility disorder that that may pose a safety risk during placement or removal of the device.
   * Gastric Mass.
   * Severe coagulopathy.
   * Taking aspirin, anti-inflammatory agents, anticoagulants or other gastric irritants and not under medical supervision.
   * Prior surgery involving the esophagus, stomach, and duodenum or bariatric surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include Obese patients (BMI 30-50 kg/m2) who have already consented to receive the Orbera365™ IGB System, who previously failed to achieve and maintain weight loss with a supervised weight-control program.
  Study subjects will also include obese and super obese patients (BMI 40 kg/m2 and above or a BMI of 35 kg/m2 with comorbidities) prior to obesity or other surgery, in order to reduce surgical risk.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Rate of Subjects with Serious Adverse Events | Up to 12 months
  The rate of subjects with serious adverse events of interest associated with the extended length of the study device in-dwell time (between 6 and 12 months) and requiringe hospitalization, endoscopic or surgical intervention, or are life-threatening. Adverse events of interest include gastric outlet obstruction, spontaneous deflation that leads to obstruction, hyperinflation, and removal complications related to airway obstruction or esophageal laceration / perforation associated with compromised balloon integrity.
Rate of Treatment Completers | Up to 12 months
  The rate of Treatment Completers that achieve ≥10% percent Total Body Weight Loss (%TBWL) at time of study removal procedure. Treatment Completer is defined as maintaining device therapy for the prescribed maximum allowed in-dwell period (up to12 months) or successfully achieving weight loss goal (e.g., at least 5% TBWL) and an early device removal for a reason other than an adverse event.

OTHER OUTCOMES:
Rate of Study Procedure-Related Adverse Events | Up to 13 months
  Continuous assessment of safety of Orbera365™ IGB System by summarizing the occurrence of study device and study procedure-related Adverse Events through 30 days post balloon removal.
Percent Total Body Weight Loss (% TBWL) at study visits through time of removal | Up to 12 months
  Percent Total Body Weight Loss (% TBWL) at study visits through time of removal (no more than 12 months).
Change in A1C | Up to 12 months
  Change in Hemoglobin A1C from baseline
Change in Insulin | Up to 12 months
  Change in Insulin from baseline
Change in Fasting Glucose | Up to 12 months
  Change in Fasting Glucose from baseline
Change in Total Cholesterol | Up to 12 months
  Change in Total Cholesterol from baseline
Change in Low-density lipoprotein (LDL) | Up to 12 months
  Change in LDL from baseline
Change in High-denisty lipoprotein (HDL) | Up to 12 months
  Change in HDL from baseline
Change in Triglycerides | Up to 12 months
  Change in Triglycerides from baseline
Change in Alanine Transaminase (ALT) | Up to 12 months
  Change in ALT from baseline
Change in Alkaline Phosphatase (ALP) | Up to 12 months
  Change in ALP from baseline
Change in Aspartate aminotransferase (AST) | Up to 12 months
  Change in AST from baseline
Change in Albumin | Up to 12 months
  Change in Albumin from baseline
Change in Direct Bilirubin | Up to 12 months
  Change in Direct Bilirubin from baseline
Change in Total Bilirubin | Up to 12 months
  Change in Total Bilirubin from baseline
Change in systolic and diastolic blood pressures | Up to 12 months
  Change in systolic and diastolic blood pressures from baseline
Changes in severity of obstructive sleep apnea (OSA) | Up to 12 months
  Changes in severity of OSA from baseline as measured by apnea-hypopnea index (AHI)
Changes in Medications for Type 2 diabetes | Up to 12 months
  Changes in Type 2 diabetes medication dose and frequency from Baseline
Changes in Hypertension Medication | Up to 12 months
  Changes in Hypertension Medication dose and frequency from baseline
Changes in Cholesterol Mediciation | Up to 12 months
  Changes in Cholesterol Medication dose and frequency from Baseline
Changes in obstructive sleep apnea (OSA) Medication and/or Medical Treatment | Up to 12 months
  Changes in OSA Medication dose and frequency and/or changes in Medical Treatment from Baseline

CONTACTS AND LOCATIONS:
Locations (5):
- OB Klinika, Prague, Czechia
- Hôpital Avicenne, Bobigny, France
- Spain (2):
  - EndoBes - Centre Medico Teknon, Barcelona
  - Dorsia Clinic, Madrid Spain, Madrid
- UHCW NHS Trust, Coventry, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: No